CLINICAL TRIAL: NCT02148185
Title: A Phase I, Open-label Study to Evaluate PK, PD, and Safety of a Single Oral Dose of MT-1303 in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Pharmacokinetics (PK), Pharmacodynamics (PD) and Safety Study of MT-1303 in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-J02
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — amiselimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MT-1303 (Experimental)
  Interventions: Drug: MT-1303

INTERVENTIONS:
Drug: MT-1303

SUMMARY:
The purpose of this study is to evaluate PK, PD and safety of a single oral dose of MT-1303 in subjects with Crohn's disease.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomised, multicenter single-dose study to evaluate PK, PD, and safety of a single oral dose of MT-1303 in subjects with moderate to severe active Crohn's disease (ileal and ileo-colonic type).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were diagnosed as Crohn's disease
* Subjects who were confirmed as ileal or ileo-colonic type by image inspection.
* Disease severity determined as either "moderate" or "severe"

Exclusion Criteria:

* Present or past history of gastrointestinal surgery which may have impact on drug absorption
* Subjects with stenosis or fistula in small intestine or colon

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of MT-1303 | 15 time points up to 29 days
Plasma concentration of MT-1303 metabolite | 15 time points up to 29 days

SECONDARY OUTCOMES:
Change from baseline in lymphocyte count after MT-1303 administration | 16 time points up to 29 days
Type of adverse events | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Mamoru Watanabe, MD, Study Director — Tokyo Medical and Dental University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (2):
- Japan (2):
  - Inverstigational site, Chūbu
  - Inverstigational site, Kanto